CLINICAL TRIAL: NCT02847923
Title: Software for Alternative Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Instituto Federal de Educação, Ciência e Tecnologia de São Paulo - IFSP (Unknown)
Responsible Party: Principal Investigator, Flavio Cezar Amate, Research Professor, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 49324115.0.0000.5497
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Speech Impairment
Keywords: Mobile Devices; Augmentative and Alternative Communication; Cerebral Palsy
MeSH Terms: conditions — Speech Disorders; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Experimental (Experimental): All the volunteers will use the software and then answer the questionnaire. They will be familiar with the software interface, performs an initial test to learn how to use the software, run a test script and answer the questionnaire.
  Interventions: Other: Presentation of alternative communication application; Other: Familiarization with the software interface; Other: Test of the software; Other: Answer the questionnaire

INTERVENTIONS:
Other: Presentation of alternative communication application — At this stage the purpose of the application is submitted, what its purpose and its features in a brief and clear manner.
Other: Familiarization with the software interface — At this stage, the volunteer will be asked to use the application by himself for a short time so that he can get acquainted and learn to use it
Other: Test of the software — Then, the volunteer is instructed to use the application following a script task that will expose a simple and fast way all the application features. These tasks have easy actions to be executed, for example: The user must communicate through the application the phrase "I want to drink water," so that he will be instructed to perform the actions to select the option and then drink the water option.
Other: Answer the questionnaire — After performing all the tasks the user replies to a questionnaire to evaluate the usability of the application after you use.

SUMMARY:
The aim of this study is evaluate a software developed for alternative communication designed for people with speech difficulties. The software was executed by 30 volunteers using mobile devices that helped to play the scenarios simulated of communication situations.

DETAILED DESCRIPTION:
Communication is a fundamental element that contributes to the development of the human being, promoting their coexistence in society. However, several factors, among them the Cerebral palsy (CP), can cause changes in muscle tone, causing injury in phono-articulatory which prevent or impair the speech production. This research aims to the development of a mobile application to promote the augmentative and alternative communication for people with CP, which adapt to the characteristics of motor limitations of these users. A mobile application was developed with pictographic resources and a voice synthesis engine, which can be customized according to the level of motor impairment and need for communication of the user. Were recruited 30 volunteers with CP who have speech difficulties and motor impairment. By means of a test script, these volunteers have used the mobile application and evaluated their usability using the questionnaire System Usability Scale (SUS), which contains 10 questions related to the ease of learning, efficiency, ease of memorization, occurrence of runtime errors of execution and level of user satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy and speech disorder

Exclusion Criteria:

* visual impairment and / or severe cognitive impairment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 15 minutes
  Questionnaire based in System Usability Scale (SUS) with 10 item questionnaire and five response options for respondents. Each response can be chosen in range: totally disagree, disagree, neither agree nor disagree, agree and totally agree.

CONTACTS AND LOCATIONS:
Overall Officials: Flávio C Amate, Dr, Principal Investigator — Núcleo de Pesquisas Tecnologicas - NPT/UMC
Locations (2):
- Brazil (2):
  - Cid Torquato, Mogi das Cruzes, São Paulo
  - Sesi Suzano, Suzano, São Paulo

IPD SHARING:
Plan to Share IPD: No